CLINICAL TRIAL: NCT03286413
Title: Comparison of Ultrasound Guided Percutaneous Microwave Ablation With Cryoablation for Breast Tumor
Brief Title: Comparison of Microwave Ablation With Cryoablation for Breast Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Prof., Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66939530yj
Record Dates: First submitted 2017-08-08; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Breast Tumor; Microwave Ablation; Cryoablation
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microwave ablation (Experimental): Microwave ablation（MWA）refers to all electromagnetic methods of inducing tumor destruction by using devices with frequencies greater than or equal to 900MHz. The rotation of dipole molecules accounts for most of the heat generated during MWA. Water molecules as dipoles attempt to continuously reorient at the same rate in microwave's oscillating electric field. As a result of microwave transmission, the water molecules flip back and forth billions of times a second. The vigorous movement of water molecules produce friction and heat, thus inducing cellular death via coagulation necrosis. The microwave unit (KY-2000, Kangyou Medical, Nanjing, China) is capable of producing 100 Watts of power at 2450 MHz.The needle antenna has a diameter of 1.6 mm (16G) and a length of 10 cm. The active tip length is 3mm and 5mm.
  Interventions: Procedure: microwave ablation
- cryoablation (Active Comparator): Clinically, cryosurgery is accomplished by placing a cryoprobe(up to 3.5 mm) through a stab incision into the tumor under ultrasound guidance.Liquid nitrogen is utilized under low operating pressure as cryogen which is controlled by the computer modulated cryogen regulator. The cryoprobe achieves rapid freezing by means of an active freeze zone at its distal tip.
  Interventions: Procedure: microwave ablation

INTERVENTIONS:
Procedure: microwave ablation — Microwave ablation and cryoablation are both thermal ablation techniques for minimally invasive treatment of breast tumor. They are performed percutaneously by ultrasound guidance.The tumor can be completely killed without injurying adjacent tissue.
  Other Names: cryoablation

SUMMARY:
The investigators will perform this study to prospectively compare the clinical outcome after percutaneous microwave ablation(MWA) and cryoablation of benign and malignant breast lesion under ultrasound (US) guidance.

DETAILED DESCRIPTION:
A total of more than 200 patients diagnosed with benign breast lesions and 50 patients with malignant breast lesions in two centers of China will be recruited in this study and underwent US-guided percutaneous MWA and cryoablation treatment. Information for each patient includes demographics; longest diameters of tumors; tumor numbers; tumor pathological type; location of tumor according to whether adjacent to skin, pectoralis, areola and papilla. Ablation variables including session, puncture, time, and power; complete ablation, complications; reduction in volume, palpability, pain and cosmetic satisfying outcomes,recurrence,survival will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* (a) the breast tumor obtained the pathological diagnosis by using core-needle biopsy; (b) for the benign lesion, continually increasing during a half year followup,with the symptoms of local pain, discomfortable or compression considered probably relating to the mass of breast; the patient with evidently psychological pressure due to the occurrence of the BBL despite clearly benignancy on imaging; (c) for the malignant lesion, with the tumor size smaller than 2cm and without other metastasis.

Exclusion Criteria:

* (a) the patients who were pregnant or breast-feeding; (b) the patients with evidence of coagulopathy or acute or severe pulmonary insufficiency or heart dysfunction; (c) the patients during menstrual period; (d) the patients referring to other therapies including surgical excision and vacuum-assisted biopsy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
volume reduce rate | 3 year
  divide the volume of ablation zone by unablated lesion volume
overall survival | 5 year

SECONDARY OUTCOMES:
local tumor progress | 5 year
  any nodular occurence adjacent to the ablation zone during the follow-up
metastasis | 5 year
  any nodular occurence keeping away from the ablation zone during the follow-up
complication | 5 year
  numbers of participants with side effect and major complications

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China